CLINICAL TRIAL: NCT00103844
Title: A Randomized Multi-Center Open Label Study of BMS-354825 vs. Imatinib Mesylate (Gleevec) 800 mg/d in Subjects With Chronic Phase Philadelphia Chromosome-Positive Chronic Myeloid Leukemia Who Have Disease That is Resistant to Imatinib at a Dose at 400 - 600 mg/d
Brief Title: Dasatinib (BMS-354835) Versus Imatinib Mesylate in Subjects With Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA180-017
Record Dates: First submitted 2005-02-15; First posted 2005-02-16 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Myeloid Leukemia; Philadelphia-Positive Myeloid Leukemia
Keywords: Chronic Phase Philadelphia chromosome Positive (Ph+) chronic myeloid leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Active Comparator
  Interventions: Drug: Dasatinib
- 2 (Experimental): Active Comparator
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, oral, 20 mg and 50mg, twice daily, up to 96 weeks
  Other Names: Sprycel; BMS-354825
  Arms: 1
Drug: Imatinib — Tablets, Oral, 400mg and 100mg, twice daily, up to 96 weeks
  Arms: 2

SUMMARY:
The primary purpose of this study is to estimate the major cytogenetic response rates of BMS-354825 and imatinib (800 mg/d) in subjects with chronic phase, Philadelphia chromosome positive, chronic myeloid leukemia (PH+ CML) with disease resistant to imatinib at a dose of 400-600 mg/d.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years of age or older.
* Subjects with Chronic Phase Ph+ CML.
* Subjects have not been treated with imatinib at a dose >600 mg/day.
* Subjects developed resistance to disease while receiving an imatinib dose 400-600 mg/day.
* Able to tolerate imatinib at the highest dose the subject had received in the past.
* Demonstrate adequate renal and hepatic function.
* Women of childbearing potential must have a negative serum or urine pregnancy test, must be using an adequate method of contraception.

Exclusion Criteria:

* Women who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period for a least 1 month before and at least 3 months after the completion of the study.
* Women using a prohibited contraceptive method.
* Women who are pregnant or breastfeeding.
* Men whose sexual partners are women who are of childbearing potential, and who are unwilling or unable to use an acceptable method to avoid pregnancy of his partner for the entire study period as outlined above.
* Prior treatment with imatinib at a dose >600 mg/day.
* Subjects who have previously identified specific BCR-ABL mutations.
* Previous diagnosis of accelerated phase or blast crisis CML.
* Intolerance to imatinib at any dose.
* Subjects who are eligible and willing to undergo transplantation during the screening period.
* Serious uncontrolled medical disorder or active infection.
* Uncontrolled or significant cardiovascular disease.
* Uncontrolled hypertension.
* Dementia or altered mental status.
* Evidence of organ dysfunction.
* Use of imatinib within 7 days.
* Use of interferon or cytarabine within 14 days.
* Use of a targeted small molecule anticancer agent within 14 days.
* Subjects taking certain medications that are accepted to have a risk of causing Torsades de Pointes.
* Subjects taking medications that irreversibly inhibit platelet function or anticoagulants.
* Prior therapy with BMS-354825.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-02; Primary Completion 2006-08 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (131):
- United States (53):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Anaheim, California
  - Local Institution, Bakersfield, California
  - Local Institution, Fullerton, California
  - Local Institution, Loma Linda, California
  - Local Institution, Los Angeles, California
  - Local Institution, Monterey Park, California
  - Local Institution, San Diego, California
  - Local Institution, Santa Barbara, California
  - Local Institution, Santa Maria, California
  - Local Institution, Stanford, California
  - Local Institution, Vallejo, California
  - Local Institution, Aurora, Colorado
  - Local Institution, Hartford, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Jacksonville, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Athens, Georgia
  - Local Institution, Atlanta, Georgia
  - Local Institution, Lawrenceville, Georgia
  - Local Institution, Tucker, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Peoria, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Kansas City, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Boston, Massachusetts
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Rochester, Minnesota
  - Local Institution, Columbia, Missouri
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Omaha, Nebraska
  - Local Institution, Hackensack, New Jersey
  - Local Institution, Morristown, New Jersey
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Cary, North Carolina
  - Local Institution, Chapel Hill, North Carolina
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Portland, Oregon
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Greenville, South Carolina
  - Local Institution, Nashville, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution, Fort Worth, Texas
  - Local Institution, Houston, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Tyler, Texas
  - Local Institution, Norfolk, Virginia
  - Local Institution, Seattle, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Vancouver, Washington
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
- Australia (5):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, St Leonards, New South Wales
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Perth, Western Australia
- Local Institution, Wein, Austria
- Belgium (6):
  - Local Institution, B-Leuven
  - Local Institution, Bruges
  - Local Institution, Brussels
  - Local Institution, Charleroi
  - Local Institution, Edegem
  - Local Institution, Yvoir
- Brazil (3):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, São Paulo, São Paulo
- Canada (4):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- China (2):
  - Local Institution, Beijing
  - Local Institution, Shanghai
- Local Institution, Aarhus, Denmark
- Local Institution, Tallinn, Estonia
- Local Institution, Helsinki, Finland
- France (7):
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (6):
  - Local Institution, Dresden
  - Local Institution, Groenkloof
  - Local Institution, Hamburg
  - Local Institution, Leipzig
  - Local Institution, Mainz
  - Local Institution, Mannheim
- Local Institution, Budapest, Hungary
- Local Institution, Dublin, Ireland
- Local Institution, Ramat Gan, Israel
- Italy (6):
  - Local Institution, Bari
  - Local Institution, Bologna
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Orbassano
  - Local Institution, Roma
- Local Institution, Trondheim, Norway
- Local Institution, Lima, Lima Province, Peru
- Local Institution, Quezon City, Philippines
- Poland (4):
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Lublin
  - Local Institution, Warsaw
- Local Institution, San Juan, Puerto Rico
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Singapore, Singapore
- South Africa (3):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Parktown, Gauteng
  - Local Institution, Soweto, Gauteng
- Local Institution, Kyunggi-Do, South Korea
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Sweden (5):
  - Local Institution, Gothenburg
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Umeå
  - Local Institution, Uppsala
- Switzerland (2):
  - Local Institution, Basel
  - Local Institution, Bellinzona
- Taiwan (2):
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- Local Institution, Bangkok, Thailand
- United Kingdom (3):
  - Local Institution, Glasglow, Central
  - Local Institution, London, Greater London
  - Local Institution, Newcastle, Tyne and Wear

REFERENCES:
- [Background] Kantarjian H, Pasquini R, Levy V, Jootar S, Holowiecki J, Hamerschlak N, Hughes T, Bleickardt E, Dejardin D, Cortes J, Shah NP. Dasatinib or high-dose imatinib for chronic-phase chronic myeloid leukemia resistant to imatinib at a dose of 400 to 600 milligrams daily: two-year follow-up of a randomized phase 2 study (START-R). Cancer. 2009 Sep 15;115(18):4136-47. doi: 10.1002/cncr.24504. PMID 19536906
- [Background] Muller MC, Cortes JE, Kim DW, Druker BJ, Erben P, Pasquini R, Branford S, Hughes TP, Radich JP, Ploughman L, Mukhopadhyay J, Hochhaus A. Dasatinib treatment of chronic-phase chronic myeloid leukemia: analysis of responses according to preexisting BCR-ABL mutations. Blood. 2009 Dec 3;114(24):4944-53. doi: 10.1182/blood-2009-04-214221. Epub 2009 Sep 24. PMID 19779040

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 166 subjects enrolled; 16 failed screening and were not treated (2 subjects were double-randomizations, 13 subjects failed inclusion criteria, 1 subject withdrew consent during screening.)
Groups:
- Dasatinib First: Dasatinib 70 mg twice a day (BID) in the first intervention period and, if intolerance to dasatinib or progression, imatinib 400 mg BID in the second intervention period (after washout period).
- Imatinib First: Imatinib 400 mg BID in the first intervention period and, if intolerance to imatinib or progression or lack of efficacy, dasatinib 70 mg BID in the second intervention period (after washout period).
Period: Overall Study
Arm/Group | Dasatinib First | Imatinib First
Started | 101 | 49
Crossed Over | 22 (22 participants from the dasatinib arm crossed over to imatinib) | 40 (40 participants from the imatinib arm crossed over the dasatinib)
Completed | 101 (Completed=no longer on treatment.Treatment continued until disease progression/intolerable toxicity.) | 49 (Completed=no longer on treatment.Treatment continued until disease progression/intolerable toxicity.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dasatinib: Dasatinib 70 mg twice a day (BID)
- Imatinib: Imatinib 400 mg BID
- Total: Total of all reporting groups
Arm/Group | Dasatinib | Imatinib | Total
Number analyzed (Participants) | 101 | 49 | 150
Age, Customized [Number; unit: participants]
  Between 21 and 45 years | 36 | 15 | 51
  Between 46 and 65 years | 48 | 28 | 76
  Between 66 and 75 years | 13 | 5 | 18
  >75 years | 4 | 1 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (13.6) | 50 (13.6) | 51 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 27 | 75
  Male | 53 | 22 | 75
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 6 | 3 | 9
  Black or African American | 2 | 1 | 3
  White | 87 | 43 | 130
  Other | 6 | 2 | 8
Eastern Cooperative Oncology Group Performance Status Scale (ECOG PS) [Number; unit: Participants] — ECOG PS: a 6-item scale to assess disease progression, daily functioning, and appropriate treatment and prognosis. Scale: 0-5, with 0=fully active, able to carry on all pre-disease performance without restriction and 5=death.
  Participants
    Score=0 (fully active) | 71 | 34 | 105
    Score=1 (ambulatory, light/sedentary work) | 27 | 12 | 39
    Score=2 (ambulatory, all selfcare, unable to work) | 0 | 0 | 0
    Score=3 (limited selfcare, some bed confinement) | 0 | 0 | 0
    Score=4 (completely disabled) | 0 | 0 | 0
    Score=5 (dead) | 0 | 0 | 0
    Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Cytogenetic Response (MCyR) at Week 12
Description: Cytogenetic response was based on the prevalence of Philadelphia chromosome positive (Ph+) metaphases among cells in metaphase on a bone marrow sample (aspirate/biopsy). MCyR was defined as Complete CyR (CCyR; 0% Ph+ cells in metaphase in bone marrow) or Partial CyR (PCyR; >0% to 35% Ph+ cells in metaphase in bone marrow).
Time Frame: Week 12
Population: All randomized subjects
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 101 | 49
Participants | 36 | 14

2. Secondary Outcome: MCyR at Any Time Prior to Crossover
Description: Cytogenetic response was based on the prevalence of Ph+ metaphases among cells in metaphase on a bone marrow sample (aspirate/biopsy). MCyR was defined as CCyR (0% Ph+ cells in metaphase in bone marrow) or PCyR (>0% to 35% Ph+ cells in metaphase in bone marrow).
Time Frame: Baseline (within 4 weeks of Day 1), every 12 weeks until crossover or off-study timepoints. Restricted to precrossover measurements.
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 101 | 49
Participants
  MCyR (CCyR + PCyR) | 54 | 16
  CCyR (0% Ph+ cells) | 44 | 9
  PCyR (>0% to 35% Ph+ cells) | 10 | 7

3. Secondary Outcome: Duration of MCyR at 12 Months and 18 Months
Description: Percentage of participants who achieved MCyR and did not progress at 12 and 18 months.
Time Frame: 12 months, 18 months
Measure: Number; unit: percentage of participants.
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 101 | 49
percentage of participants.
  12 months | 92 | 74
  18 months | 90 | 74

4. Secondary Outcome: Duration of MCyR at 24 Months
Description: Percentage of participants who achieved MCyR and did not progress at 24 months.
Time Frame: 24 Months
Population: In the imatinib group, the 24 months timepoint was beyond the maximum observed time.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 101 | 0
Percentage of Participants | 90 |

5. Secondary Outcome: Time to MCyR Prior to Crossover
Description: Median time from first dosing date to date of MCyR
Time Frame: Baseline (within 4 weeks of Day 1), every 12 weeks, at crossover or off-study timepoints; restricted to precrossover measurements.
Population: Population consists of the number of responders in each treatment group
Measure: Median (Full Range); unit: months
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 54 | 16
months | 2.8 [0.7 to 19.3] | 2.8 [2.4 to 5.7]

6. Secondary Outcome: Complete Hematologic Response (CHR) at Any Time Prior to Crossover
Description: Participants achieving CHR prior to crossover. CHR=all of the following criteria: white blood cell count ≤ institutional upper limit of normal; platelets < 450,000/mm³; no blasts or promyelocytes in peripheral blood; < 5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils ≤ 20%; no extramedullary involvement. Confirmed CHR is defined as CHR maintained at least 4 weeks after first documented at ≥ Day 14. Failure to maintain criteria of CHR was defined by 2 or more consecutive records of non-response.
Time Frame: Baseline (within 4 weeks of Day 1), weekly until Week 12 and then every 12 weeks until crossover or off-study; restricted to precrossover measurements.
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 101 | 49
Participants | 94 | 40

7. Secondary Outcome: Duration of Complete Hematologic Response (CHR)
Description: Percentage of participants who achieved CHR and did not progress at specified time points. CHR=all of the following criteria: white blood cell count ≤ institutional upper limit of normal; platelets < 450,000/mm³; no blasts or promyelocytes in peripheral blood; < 5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils ≤ 20%; no extramedullary involvement. Confirmed CHR is defined as CHR maintained at least 4 weeks after first documented at ≥ Day 14. Failure to maintain criteria of CHR was defined by 2 or more consecutive records of non-response.
Time Frame: 12 months, 24 months
Population: Number of participants achieving CHR in each treatment group
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 94 | 40
percentage of participants
  12 months | 92 | 82
  24 months | 84 | 73

8. Secondary Outcome: Time to CHR Prior to Crossover
Description: Median time from first dosing date to date of CHR. CHR=all of the following criteria: white blood cell count ≤ institutional upper limit of normal; platelets < 450,000/mm³; no blasts or promyelocytes in peripheral blood; < 5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils ≤ 20%; no extramedullary involvement. Confirmed CHR is defined as CHR maintained at least 4 weeks after first documented at ≥ Day 14. Failure to maintain criteria of CHR was defined by 2 or more consecutive records of non-response.
Time Frame: Baseline (within 4 weeks of Day 1), weekly until Week 12, then every 12 weeks until crossover or off-study; restricted to precrossover measurements.
Population: Number of participants achieving CHR in each treatment group
Measure: Median (Full Range); unit: weeks
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 94 | 40
weeks | 2.1 [2 to 15.9] | 2.1 [2 to 6.1]

9. Secondary Outcome: Major Molecular Response (MMR)
Description: Number of participants Achieving MMR. MMR is defined as ≤3 log reduction (ie, international ratio ≤0.1), in BCR-ABL levels from the standardized baseline value of BCR-ABL: Control Gene ratio. The international ratio is obtained by multiplying BCR-ABL: Control gene ratio by the lab-specific conversion factor.
Time Frame: Pretreatment, then after every 4 weeks for 12 weeks, then after every 12 week period out to 2 years; restricted to precrossover measurements.
Population: Participants assessed for MMR only
Measure: Number; unit: participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 99 | 45
participants | 29 | 6

10. Secondary Outcome: CHR After Crossover
Description: Participants achieving CHR after crossover. CHR=all of the following criteria: white blood cell count ≤ institutional upper limit of normal; platelets < 450,000/mm³; no blasts or promyelocytes in peripheral blood; < 5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils ≤ 20%; no extramedullary involvement. Confirmed CHR is defined as CHR maintained at least 4 weeks after first documented at ≥ Day 14. Failure to maintain criteria of CHR was defined by 2 or more consecutive records of non-response.
Time Frame: Weekly for 12 weeks, then after every 12 week period out to 2 years; restricted to postcrossover measurements.
Population: Participants evaluable for response after crossover
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 39 | 20
Participants | 37 | 13

11. Secondary Outcome: Cytogenetic Response After Crossover
Description: Cytogenetic response was based on the prevalence of Ph+ metaphases among cells in metaphase on a bone marrow sample (aspirate/biopsy). MCyR was defined as Complete CyR (0% Ph+ cells in metaphase in bone marrow) or Partial CyR (>0% to 35% Ph+ cells in metaphase in bone marrow).
Time Frame: every 12 week period out to 2 years and off-study timepoints; restricted to postcrossover measurements
Population: Participants evaluable for after crossover response
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 39 | 20
Participants
  Major Cytogenetic Response (MCyR) | 19 | 3
  Complete Cytogenetic Response (CCyR) | 15 | 0
  Partial Cytogenetic Response (PCyR) | 4 | 3

12. Secondary Outcome: Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths and Hematologic Toxicities Prior to Crossover
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition regardless of causal relationship with treatment. SAE=any untoward medical occurrence at any dose that: results in death; is life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability; is cancer; is congenital anomaly/birth defect; results in drug dependency/abuse; is an important medical event. Graded by National Cancer Institute Common Terminology Criteria for Adverse Events v3.0. (1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death)
Time Frame: Continuously from baseline through 2 years
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 101 | 49
Participants
  Any Adverse Event (AE) | 100 | 45
  Grade 3-4 AEs | 67 | 21
  Drug-related AEs | 94 | 44
  Drug-related Grade 3-4 AEs | 62 | 19
  Death within 30 days of last dose | 1 | 0
  Drug-related Serious AEs | 28 | 3
  AEs leading to discontinuation | 23 | 10
  Fluid Retention AEs - Overall | 39 | 21
  Fluid Retention AEs - Superficial Edema | 20 | 21
  Fluid Retention AEs - Pleural Effusion | 25 | 0
  Fluid Retention AEs - Other | 9 | 0
  Grade 3-4 Hematologic Toxicity - Anemia | 20 | 4
  Grade 3-4 Hematologic Toxicity - Thrombocytopenia | 58 | 7
  Grade 3-4 Hematologic Toxicity - Neutropenia | 64 | 19
  Grade 3-4 Hematologic Toxicity - Leukopenia | 24 | 8

13. Secondary Outcome: Health-Related Quality of Life Prior to Crossover
Description: Health-related quality of life as measured by Functional Assessment of Cancer Therapy-General (FACT-G). FACT-G=27 questions in 4 domains: physical, social/family, emotional, & functional well-being (PWB, SWB, EWB, FWB). Higher scores=better health-related quality of life. Total Score change of 7 or more=minimal clinical important change; PWB, EWB, & FWB score change of 3 or more, & SWB score change of 2 or more=minimal clinical important change.
Time Frame: Every 4 weeks for the first 24 weeks, then every 12 weeks for the remainder of treatment. Last questionnaire was to be completed at first follow-up visit after off-study date.
Population: Since single-arm quality-of-life data are not interpretable in a non-comparative trial, these data were not analyzed.
Measure: Number; unit: Units on a Scale
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Blood Sample Collection for Pharmacokinetic (PK) Analysis of Dasatinib
Description: Number of participants from which blood samples were collected for population PK studies.
Time Frame: Day 8: pretreatment trough sample, a sample between 30 minutes and 3 hours following treatment, a sample between 5 and 8 hours following treatment, and a sample at 12 hours, prior to the next dose.
Population: Blood samples that were to contribute to PK modeling were collected from 78 participants,to be included in separate population PK analyses. Although blood sample collection was listed as a secondary endpoint, no study-specific PK analyses were planned for this report.
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 78
participants | 78

ADVERSE EVENTS:
Arm/Group | DASATINIB | IMATINIB
Serious Adverse Events (participants affected / at risk) | 43/101 | 4/49
Other Adverse Events (participants affected / at risk) | 99/101 | 43/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DASATINIB (N=101) | IMATINIB (N=49)
CATARACT (Eye disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 | 0
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
HEPATIC LESION (Hepatobiliary disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
ANORECTAL DISORDER (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
MUMPS (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 2 | 0
PNEUMONIA (Infections and infestations) | 7 | 0
CELLULITIS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 | 0
UTERINE DILATION AND CURETTAGE (Surgical and medical procedures) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 0
ANAEMIA (Blood and lymphatic system disorders) | 3 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 1
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 10 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DEATH (General disorders) | 1 | 0
PYREXIA (General disorders) | 5 | 0
CHEST DISCOMFORT (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 0
ANAL CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLAST CRISIS IN MYELOGENOUS LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DASATINIB (N=101) | IMATINIB (N=49)
EYE OEDEMA (Eye disorders) | 1 | 3
EYELID OEDEMA (Eye disorders) | 3 | 4
CONJUNCTIVITIS (Eye disorders) | 6 | 2
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 6 | 0
WEIGHT DECREASED (Investigations) | 27 | 4
WEIGHT INCREASED (Investigations) | 14 | 8
HYPERTENSION (Vascular disorders) | 9 | 0
INSOMNIA (Psychiatric disorders) | 9 | 3
HEADACHE (Nervous system disorders) | 46 | 6
DIZZINESS (Nervous system disorders) | 18 | 3
NAUSEA (Gastrointestinal disorders) | 32 | 19
VOMITING (Gastrointestinal disorders) | 18 | 13
DIARRHOEA (Gastrointestinal disorders) | 48 | 14
DYSPEPSIA (Gastrointestinal disorders) | 12 | 4
GASTRITIS (Gastrointestinal disorders) | 9 | 1
TOOTHACHE (Gastrointestinal disorders) | 9 | 1
STOMATITIS (Gastrointestinal disorders) | 6 | 2
CONSTIPATION (Gastrointestinal disorders) | 9 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 16 | 5
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 7 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 15 | 0
RHINITIS (Infections and infestations) | 9 | 0
PNEUMONIA (Infections and infestations) | 7 | 0
SINUSITIS (Infections and infestations) | 7 | 1
BRONCHITIS (Infections and infestations) | 10 | 2
ORAL HERPES (Infections and infestations) | 8 | 2
PHARYNGITIS (Infections and infestations) | 9 | 1
GASTROENTERITIS (Infections and infestations) | 8 | 0
NASOPHARYNGITIS (Infections and infestations) | 12 | 2
URINARY TRACT INFECTION (Infections and infestations) | 6 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 | 7
ANOREXIA (Metabolism and nutrition disorders) | 23 | 4
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 3
ANAEMIA (Blood and lymphatic system disorders) | 8 | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 22 | 8
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 22 | 5
RASH (Skin and subcutaneous tissue disorders) | 30 | 9
ALOPECIA (Skin and subcutaneous tissue disorders) | 11 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 12 | 1
PETECHIAE (Skin and subcutaneous tissue disorders) | 6 | 2
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 2 | 3
PERIORBITAL OEDEMA (Skin and subcutaneous tissue disorders) | 3 | 4
BREAST PAIN (Reproductive system and breast disorders) | 7 | 0
CONTUSION (Injury, poisoning and procedural complications) | 7 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 13 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 13 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 17 | 8
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 | 8
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 20 | 6
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 12 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 29 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 25 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 22 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 12 | 2
PAIN (General disorders) | 5 | 3
CHILLS (General disorders) | 6 | 4
FATIGUE (General disorders) | 46 | 12
PYREXIA (General disorders) | 32 | 8
ASTHENIA (General disorders) | 19 | 3
CHEST PAIN (General disorders) | 8 | 0
FACE OEDEMA (General disorders) | 6 | 7
FEELING COLD (General disorders) | 3 | 3
OEDEMA PERIPHERAL (General disorders) | 18 | 10
INFLUENZA LIKE ILLNESS (General disorders) | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.